CLINICAL TRIAL: NCT01519544
Title: Treatment of High-altitude Sleep Disturbance: A Double-blind Comparison of Temazepam Versus Acetazolamide.
Brief Title: Comparison of Temazepam and Acetazolamide to Treat Difficulty Sleeping at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, N. Stuart Harris MD MFA, Director, MGH Wilderness Medicine Fellowship; Chief, Division of Wilderness Medicine, Department of Emergency Medicine, Massachusetts General Hospital; Assistant Professor of Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P000017
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: High-altitude Sleep Disturbance
Keywords: Sleep; High Altitude; High-altitude Sleep Disturbance; Acute Mountain Sickness; Difficulty Sleeping at High Altitude; Periodic Breathing; Actigraphy; Acetazolamide; Temazepam; Groningen Sleep Quality Questionnaire survey; Stanford Sleepiness Scale; Lake Louise Acute Mountain Sickness Score
MeSH Terms: conditions — Altitude Sickness | interventions — Temazepam; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temazepam (Active Comparator): 50 subjects are instructed to take 7.5mg temazepam by mouth prior to going to sleep for one night only.
  Interventions: Drug: Temazepam
- Acetazolamide (Active Comparator): 50 subjects are instructed to take 125mg of acetazolamide by mouth prior to going to sleep one night only.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Temazepam — Temazepam 7.5mg capsule to be taken by mouth at bedtime for one night only.
  Other Names: Restoril
  Arms: Temazepam
Drug: Acetazolamide — Take Acetazolamide 125mg tablet by mouth at bedtime for one night only.
  Other Names: Diamox
  Arms: Acetazolamide

SUMMARY:
More than 70% of visitors to high altitude suffer poor sleep. The present study seeks to answer the question: Which medication is associated with better sleep at high altitude: temazepam or acetazolamide? The investigators hypothesis is that one medication will be associated with higher subjective sleep scores than the other. The study will compare the sleep quality of 100 subjects as they take either temazepam or acetazolamide during a visit to high altitude.

DETAILED DESCRIPTION:
Difficulty sleeping is very common with acute high altitude exposure. Sleep disturbances were reported by more than 70% of participants in acute mountain sickness pharmacologic treatment trials. Difficulty sleeping is one of the primary complaints of visitors to high altitude and some authors consider difficulty sleeping to be nearly universal at high altitudes. Acetazolamide, temazepam, zolpidem and zaleplon are all effective and safe in treating the acute insomnia of high altitude. No head-to-head trials have been performed to determine the best drug class for treatment of high altitude sleep disturbances. The purpose of this study is to compare temazepam and acetazolamide in the treatment of high altitude sleep disturbances. Such knowledge will benefit the hundreds of thousands of visitors to areas of high altitude throughout the world.

The study will be a convenience sample of 100 trekkers in Manang, Nepal (elevation 11,500 feet). The study will only enroll trekkers who have gained more than 200 meters (650 feet) over the preceding 24 hours. Subject enrollment will take place from March 1, 2012, through May 30, 2012. One hundred subjects will be enrolled.

All subjects will complete the study in Manang, Nepal. Once an individual decides to enroll in the study, they will be instructed on the risks of the study and informed consent will be obtained. Eligibility to participate will be verified.

Each subject will be randomly assigned to take 125 mg of acetazolamide or 7.5 mg of temazepam by mouth immediately prior to going to bed. Each subject will only take one dose of the medication as part of the trial. Subjects will wear a pulse oximeter and an actigraph to bed. An actigraph is an accelerometer that is worn like a wrist watch. Actigraphs can sense and record movement and for this reason are often used in sleep studies to help measure sleep duration and quality.

Study participants will keep a sleep log and will be asked to complete a Groningen Sleep Quality Questionnaire Survey and Lake Louise Acute Mountain Sickness questionnaire. Subjects will also complete a Stanford Sleepiness Scale every hour for eight hours.

Through both objective and subjective measurement of sleep quality, this study is designed to determine which medication is associated with improved sleep at high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Trekkers on the Annapurna circuit
* Must be in the process of ascent (> 200 meters over the previous 24 hours)
* Must be willing to stay 2 nights in Manang, Nepal
* Healthy adults, age 18-65
* Self-report of new difficulty sleeping over the previous two days

Exclusion Criteria:

* Recent (< 2 weeks) high altitude exposure (higher than 11, 500 feet or 3500 meters)
* Current acute illness
* Moderate to Severe Acute Mountain Sickness (Lake Louise AMS score > 4)
* High Altitude Cerebral Edema
* High Altitude Pulmonary Edema
* Any pre-existing sleep disorders or sleep related condition including obstructive sleep apnea, morbid obesity (BMI > 40), restless leg syndrome, etc.
* Any lung disease or condition affecting the lungs, including chronic obstructive pulmonary disease, asthma, cystic fibrosis, etc.
* Congestive heart failure, pulmonary hypertension, or cardiomyopathy
* Current oxygen use
* Kidney disease
* Liver disease
* Pregnancy or breast feeding
* Seizure disorder or other neurologic disorder
* Glaucoma
* Sulfa allergy
* Acetazolamide allergy
* Benzodiazepine allergy
* Temazepam allergy
* Currently on acetazolamide
* Currently taking any benzodiazepines
* Current medical treatment with any of the following: antidepressants, neuroleptics, anxiolytics, H1 antihistamines, barbiturates or hypnotics (including benzodiazepines or any other sleep aids).
* Major psychiatric diagnosis (depression, anxiety, schizophrenia)
* Recreational drug use
* Caffeine con¬sumption > 3 cups of coffee/day
* Alcohol consumption > 1 drink/day
* Mental Retardation or Developmental Disabilities
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Global assessment of sleep quality using a 100mm visual analog scale | 1 day
  The morning after taking the study medication, subjects will be asked: How would you rate last night's sleep quality? They will mark their answer on a 100mm visual analog scale with 0mm representing 'worst night of sleep ever' and 100mm representing 'best night of sleep ever'.
The Groningen Sleep Quality Questionnaire survey | 1 day
  The Groningen Sleep Quality Questionnaire survey includes fifteen questions that describe sleep onset, sleep quality, awakenings, sleep duration, and wake up quality. Survey is completed by the subject.

SECONDARY OUTCOMES:
Sleep Onset Latency | 1 day
  The amount of time it takes the subject to fall asleep. Reported by the subject.
Total Sleep Duration | 1 day
  The total amount of time that the subject slept. Recorded by the subject.
Time in Bed | 1 day
  The amount of time the subject spent in bed. Recorded by the subject.
Number of Awakenings | 1 day
  The number of times the subject woke up from sleep. Recorded by the subject.
Number of Awakenings to Urinate | 1 day
  Number of time the subject woke up from sleep to use the restroom. Recorded by the subject.
Wake Time After Sleep Onset | 1 day
  Amount of time the subject spent awake after falling asleep. Recorded by the subject.
Terminal Wakefulness | 1 day
  The amount of time the subject spends in bed after waking up for the last time. Reported by the subject.
Global assessment of sleep depth | 1 day
  Subjects will be asked to rate the depth of sleep on a 100mm visual analog scales.
Global assessment of drowsiness | 1 day
  Subjects will be asked to assess their daytime drowsiness on a 100mm visual analog scale.
Stanford Sleepiness Scale scores | 1 day
  During each of the eight hours after waking up, subjects will be asked to complete a Stanford Sleepiness Scale to measure how sleepy they are.
Lake Louis Acute Mountain Sickness delta score | 1 day
  Subjects will be asked to fill out a Lake Louise Acute Mountain Sickness score at the beginning and end of study participation. The Lake Louise Acute Mountain Sickness score reflects on the severity of Acute Mountain Sickness being experienced by the subject. Scores consistent moderate or severe Acute Mountain Sickness will exclude subjects from participation in the study.
Mean O2 Saturation | 1 day
  Study subjects will wear a pulse oximeter during the night that will record their oxygen saturation.
Proportion of time in periodic breathing | 1 day
  Visitors to high altitude experience periodic breathing (alternating periods of increased and decreased respiratory rate) as the human body adjusts to the hypoxemia of high altitude. Both temazepam and acetazolamide have been shown to improve periodic breathing. Subjects will wear pulse oximeters. Data from the pulse oximeters will be used to calculate the amount of time that subjects spend in periodic breathing.
Number of desaturation events per hour | 1 day
  Due to the periodic breathing that occurs at high altitude, there are frequent oxygen desaturations during sleep. Subjects will wear a pulse oximeter to determine how many time they experience a decline in their oxygen saturation during the night.
Number of awakenings per hour | 1 day
  Subjects will wear an actigraph while they sleep. Actigraphs are small wristwatch-like devices that measure subtle movements while a subject is asleep. These movements are used to objectively describe awake and asleep periods.
Sleep Efficiency | 1 day
  Subjects will wear an actigraph when they sleep. Actigraphs are small wristwatch-like devices that measure the subtle movements of a subject during the night and help objectively determine awake and asleep periods. Using data from the actigraph, one may calculate what percent of the night the subject was asleep (sleep efficiency).

CONTACTS AND LOCATIONS:
Overall Officials: Norman S Harris, MD, MFA, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Himalayan Rescue Location clinic in Manang, Manang, District of Manang, Nepal

REFERENCES:
- [Background] Larson EB, Roach RC, Schoene RB, Hornbein TF. Acute mountain sickness and acetazolamide. Clinical efficacy and effect on ventilation. JAMA. 1982 Jul 16;248(3):328-32. PMID 7045433
- [Background] Ellsworth AJ, Larson EB, Strickland D. A randomized trial of dexamethasone and acetazolamide for acute mountain sickness prophylaxis. Am J Med. 1987 Dec;83(6):1024-30. doi: 10.1016/0002-9343(87)90937-5. PMID 3332564
- [Background] Honigman B, Theis MK, Koziol-McLain J, Roach R, Yip R, Houston C, Moore LG, Pearce P. Acute mountain sickness in a general tourist population at moderate altitudes. Ann Intern Med. 1993 Apr 15;118(8):587-92. doi: 10.7326/0003-4819-118-8-199304150-00003. PMID 8452324
- [Background] Forwand SA, Landowne M, Follansbee JN, Hansen JE. Effect of acetazolamide on acute mountain sickness. N Engl J Med. 1968 Oct 17;279(16):839-45. doi: 10.1056/NEJM196810172791601. No abstract available. PMID 4877992
- [Background] Dubowitz G. Effect of temazepam on oxygen saturation and sleep quality at high altitude: randomised placebo controlled crossover trial. BMJ. 1998 Feb 21;316(7131):587-9. doi: 10.1136/bmj.316.7131.587. PMID 9518909
- [Background] Nickol AH, Leverment J, Richards P, Seal P, Harris GA, Cleland J, Dubowitz G, Collier DJ, Milledge J, Stradling JR, Morrell MJ. Temazepam at high altitude reduces periodic breathing without impairing next-day performance: a randomized cross-over double-blind study. J Sleep Res. 2006 Dec;15(4):445-54. doi: 10.1111/j.1365-2869.2006.00558.x. PMID 17118102
- [Background] Beaumont M, Batejat D, Coste O, Van Beers P, Colas A, Clere JM, Pierard C. Effects of zolpidem and zaleplon on sleep, respiratory patterns and performance at a simulated altitude of 4,000 m. Neuropsychobiology. 2004;49(3):154-62. doi: 10.1159/000076723. PMID 15034230
- [Background] Beaumont M, Batejat D, Pierard C, Van Beers P, Philippe M, Leger D, Savourey G, Jouanin JC. Zaleplon and zolpidem objectively alleviate sleep disturbances in mountaineers at a 3,613 meter altitude. Sleep. 2007 Nov;30(11):1527-33. doi: 10.1093/sleep/30.11.1527. PMID 18041485
- [Background] Sharma A, Dewan VK. A Case Report of Zolpidem-Induced Somnambulism. Prim Care Companion J Clin Psychiatry. 2005;7(2):74. doi: 10.4088/pcc.v07n0207a. No abstract available. PMID 15841201
- [Background] Yang W, Dollear M, Muthukrishnan SR. One rare side effect of zolpidem--sleepwalking: a case report. Arch Phys Med Rehabil. 2005 Jun;86(6):1265-6. doi: 10.1016/j.apmr.2004.11.022. PMID 15954071
- [Background] Auerbach, Paul S. Wilderness Medicine, 5th ed. Mosby, Phidelphia. Pages 4-8. 2007.
- [Background] Luks AM. Which medications are safe and effective for improving sleep at high altitude? High Alt Med Biol. 2008 Fall;9(3):195-8. doi: 10.1089/ham.2008.1025. PMID 18800955
- [Background] Sutton JR, Gray GW, Houston CS, Powles AC. Effects of duration at altitude and acetazolamide on ventilation and oxygenation during sleep. Sleep. 1980;3(3-4):455-64. doi: 10.1093/sleep/3.3-4.455. No abstract available. PMID 7221351
- [Background] Sutton JR, Houston CS, Mansell AL, McFadden MD, Hackett PM, Rigg JR, Powles AC. Effect of acetazolamide on hypoxemia during sleep at high altitude. N Engl J Med. 1979 Dec 13;301(24):1329-31. doi: 10.1056/NEJM197912133012406. No abstract available. PMID 503151
- [Background] Hackett PH, Roach RC, Harrison GL, Schoene RB, Mills WJ Jr. Respiratory stimulants and sleep periodic breathing at high altitude. Almitrine versus acetazolamide. Am Rev Respir Dis. 1987 Apr;135(4):896-8. doi: 10.1164/arrd.1987.135.4.896. PMID 3565935
- [Background] Fischer R, Lang SM, Leitl M, Thiere M, Steiner U, Huber RM. Theophylline and acetazolamide reduce sleep-disordered breathing at high altitude. Eur Respir J. 2004 Jan;23(1):47-52. doi: 10.1183/09031936.03.00113102. PMID 14738230
- [Background] Nicholson AN, Smith PA, Stone BM, Bradwell AR, Coote JH. Altitude insomnia: studies during an expedition to the Himalayas. Sleep. 1988 Aug;11(4):354-61. doi: 10.1093/sleep/11.4.354. PMID 2905069
- [Background] Bradwell AR, Coote JH, Smith P, et al. (1987) The effect of temazepam and Diamox on nocturnal hypoxia at altitude [abstract]. In: Sutton J.R., Houston C.S., Coates G., ed. Hypoxia and Cold, New York: Praeger; 1987: P543.
- [Background] Strom BL, Schinnar R, Apter AJ, Margolis DJ, Lautenbach E, Hennessy S, Bilker WB, Pettitt D. Absence of cross-reactivity between sulfonamide antibiotics and sulfonamide nonantibiotics. N Engl J Med. 2003 Oct 23;349(17):1628-35. doi: 10.1056/NEJMoa022963. PMID 14573734
- [Background] Roggla G, Moser B, Roggla M. Effect of temazepam on ventilatory response at moderate altitude. BMJ. 2000 Jan 1;320(7226):56. No abstract available. PMID 10617541
- [Background] Hackett PH, Roach RC. High-altitude illness. N Engl J Med. 2001 Jul 12;345(2):107-14. doi: 10.1056/NEJM200107123450206. No abstract available. PMID 11450659
- [Background] Basnyat B, Murdoch DR. High-altitude illness. Lancet. 2003 Jun 7;361(9373):1967-74. doi: 10.1016/S0140-6736(03)13591-X. PMID 12801752
- [Background] Jafarian S, Gorouhi F, Taghva A, Lotfi J. High-altitude sleep disturbance: results of the Groningen Sleep Quality Questionnaire survey. Sleep Med. 2008 May;9(4):446-9. doi: 10.1016/j.sleep.2007.06.017. Epub 2007 Sep 14. PMID 17869574
- [Background] Weil JV. Sleep at high altitude. High Alt Med Biol. 2004 Summer;5(2):180-9. doi: 10.1089/1527029041352162. PMID 15265339
- [Background] Jones JE, Muza SR, Fulco CS, Beidleman BA, Tapia ML, Cymerman A. Intermittent hypoxic exposure does not improve sleep at 4300 m. High Alt Med Biol. 2008 Winter;9(4):281-7. doi: 10.1089/ham.2008.1039. PMID 19115911
- [Background] Cole RJ, Kripke DF, Gruen W, Mullaney DJ, Gillin JC. Automatic sleep/wake identification from wrist activity. Sleep. 1992 Oct;15(5):461-9. doi: 10.1093/sleep/15.5.461. PMID 1455130
- [Background] Coffield TG, Tryon WW. Construct validation of actigraphic sleep measures in hospitalized depressed patients. Behav Sleep Med. 2004;2(1):24-40. doi: 10.1207/s15402010bsm0201_3. PMID 15600222
- [Background] Hackett P. and Olez O. (1992). The Lake Louise consensus on the definition and qualification of altitude illness. In: J. Sutton, G. Coates and C. Houston (Eds) Hypoxia and mountain medicine. Queen City Press, Burlington, 1992: 327-330.
- [Background] Mulder-Hajonides van der Meulen WREH, Wijnberg J.R., Hollander J.J., De Diana I.P.F. and van den Hoofdakker R.H. (1980) Measurement of subjective sleep quality. Eur. Sleep Res. Soc. Abstr. 5:98.
- [Background] Meesters Y, Jansen JH, Lambers PA, Bouhuys AL, Beersma DG, van den Hoofdakker RH. Morning and evening light treatment of seasonal affective disorder: response, relapse and prediction. J Affect Disord. 1993 Jul;28(3):165-77. doi: 10.1016/0165-0327(93)90102-p. PMID 8408979
- [Background] Meijman T.F., Thunnissen M.J., de Vries-Griever A.G.H. (1990) The after-effects of a prolonged period of day-sleep on subjective sleep quality. Work Stress. 4:65-70.
- [Background] Nussbaumer-Ochsner Y, Latshang TD, Ulrich S, Kohler M, Thurnheer R, Bloch KE. Patients with obstructive sleep apnea syndrome benefit from acetazolamide during an altitude sojourn: a randomized, placebo-controlled, double-blind trial. Chest. 2012 Jan;141(1):131-138. doi: 10.1378/chest.11-0375. Epub 2011 Jun 9. PMID 21659435
- [Background] Vallieres A, Morin CM. Actigraphy in the assessment of insomnia. Sleep. 2003 Nov 1;26(7):902-6. doi: 10.1093/sleep/26.7.902. PMID 14655927
- [Background] Sadeh A. The role and validity of actigraphy in sleep medicine: an update. Sleep Med Rev. 2011 Aug;15(4):259-67. doi: 10.1016/j.smrv.2010.10.001. Epub 2011 Jan 14. PMID 21237680
- [Background] Sadeh A, Hauri PJ, Kripke DF, Lavie P. The role of actigraphy in the evaluation of sleep disorders. Sleep. 1995 May;18(4):288-302. doi: 10.1093/sleep/18.4.288. PMID 7618029
- [Background] Sadeh A, Sharkey KM, Carskadon MA. Activity-based sleep-wake identification: an empirical test of methodological issues. Sleep. 1994 Apr;17(3):201-7. doi: 10.1093/sleep/17.3.201. PMID 7939118
- [Background] Jean-Louis G, Kripke DF, Mason WJ, Elliott JA, Youngstedt SD. Sleep estimation from wrist movement quantified by different actigraphic modalities. J Neurosci Methods. 2001 Feb 15;105(2):185-91. doi: 10.1016/s0165-0270(00)00364-2. PMID 11275275
- [Background] Lichstein KL, Stone KC, Donaldson J, Nau SD, Soeffing JP, Murray D, Lester KW, Aguillard RN. Actigraphy validation with insomnia. Sleep. 2006 Feb;29(2):232-9. PMID 16494091
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003
- [Background] Kryger M.H., Roth T. and Dement W.C. (2011). Chapters 143 and 147. Principles and Practice of Sleep Medicine, 5th ed. Saunders, St. Louis, 2011.
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Nussbaumer-Ochsner Y, Schuepfer N, Siebenmann C, Maggiorini M, Bloch KE. High altitude sleep disturbances monitored by actigraphy and polysomnography. High Alt Med Biol. 2011 Fall;12(3):229-36. doi: 10.1089/ham.2010.1073. PMID 21962066
- [Background] Erman MK, Zammit G, Rubens R, Schaefer K, Wessel T, Amato D, Caron J, Walsh JK. A polysomnographic placebo-controlled evaluation of the efficacy and safety of eszopiclone relative to placebo and zolpidem in the treatment of primary insomnia. J Clin Sleep Med. 2008 Jun 15;4(3):229-34. PMID 18595435
- [Background] Zammit GK, McNabb LJ, Caron J, Amato DA, Roth T. Efficacy and safety of eszopiclone across 6-weeks of treatment for primary insomnia. Curr Med Res Opin. 2004 Dec;20(12):1979-91. doi: 10.1185/174234304x15174. PMID 15701215